CLINICAL TRIAL: NCT02629133
Title: Computer-Based Intervention for Battered Sheltered Women With Substance Use Randomized Trial
Brief Title: Intervention for Battered Sheltered Women With Substance Use Randomized Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Caron Zlotnick, Director of Behavioral Medicine Research, Women and Infants Hospital of Rhode Island
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 792696; R34DA038770-01A1 (NIH)
Record Dates: First submitted 2015-12-02; First posted 2015-12-14 (Estimated); Results first posted 2020-04-08 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Intimate Partner Violence
Keywords: Intimate Partner Violence; Sheltered Battered Women; Substance Use
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SHE Program (Experimental): Participants received a 50 minute intervention on the computer immediately after their baseline assessment and a 15 minute "booster" session on the computer within 2 weeks after the intervention. There was also a 3 and 6 month follow-up after completion of the SHE program.
  Interventions: Behavioral: SHE Program
- Control Condition (No Intervention): Control condition consisted of a series of questions regarding television show preferences and viewing a brief series of videos of popular entertainers/shows, with subsequent requests for rating of subjective preference. Participants in this condition completed a baseline assessment as well as a television show booster and a follow-up assessment 3 and 6 months later.

INTERVENTIONS:
Behavioral: SHE Program — The SHE program is specifically tailored, innovative and relevant to diverse, racial, and ethnic sheltered, battered women in a number of ways including the images and content used in the intervention. It is also tailored to participants' alcohol or substance use status, and designed to reach participants across levels of motivation for change. The content of SHE is theory-driven, consistent with the motivational interviewing model of behavior, and consistent with the literature on effective interventions that address IPV and substance use.
  Arms: SHE Program

SUMMARY:
This study developed and assessed an innovative, high-reach, easily implementable, low-cost computer-delivered intervention (Safe and Healthy Experiences; The SHE Program) that addresses known barriers in early identification and intervention with sheltered battered women with IPV (intimate partner violence) and substance use.

DETAILED DESCRIPTION:
Intimate partner violence (IPV) and substance use are significant and interconnected public health problems facing women. For battered women, the presence of substance use increases the risk of revictimization and the risk of more severe abuse. Battered women's shelters provide emergency shelter to approximately 300,000 women and children each year. A prime time to intervene with battered women might be when they enter a shelter and have already initiated a change in their lives. A shelter-based intervention for battered women that addresses substance use problems might reduce the risk of substance use, reduce the risk of future IPV, and improve utilization of substance use treatment and community resources. The objective of this R34 Award was to develop and assess an innovative, easily implementable, low-cost, computer-delivered intervention, the SHE Program (Safe and Healthy Experiences) that addresses known barriers in early identification and intervention for battered sheltered women with substance use issues. SHE is based on motivational interviewing (MI) a well-defined intervention strategy that has yielded particularly promising results in a range of clinical issues and a range of patient populations, including substance using women. MI is consistent with an empowerment model, which is a highly recommended intervention model for victimized women. The R34 had two distinct phases to assess the SHE Program with battered sheltered women with substance use issues. During the Development Phase, the research team conducted focus groups and developed the intervention to meet the needs of our target group, developed the software for the computer-delivered intervention, and conducted an open trial with 10 participants. During the Pilot Study Phase, the investigators conducted a two-group, randomized controlled study with a sample of 50 battered sheltered women who reported substance use difficulties within the last three months, which provides the necessary groundwork to examine the efficacy of the SHE Program in a future, large clinical trial. The SHE Program was found to be feasible, acceptable and efficacious in improving outcomes for our vulnerable target population. The program has the potential to be widely disseminated while maintaining treatment fidelity across battered women shelters and may hold promise for IPV populations with substance use difficulties in other settings.

ELIGIBILITY:
Inclusion Criteria:

* Women who are 18 or older, residents of a battered women's shelter, who are at risk substance users within the last 3 months as determined by the screener, the NIDA-Modified ASSIST, and endorse IPV within the last 3 months as determined by the screener, the WAST (Woman Abuse Screening Tool)

Exclusion Criteria:

* Inability to provide informed consent (e.g., due to florid psychosis or other clear cognitive impairment)
* Inability to understand English

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-03; Primary Completion 2018-12 (Actual); Study Completion 2019-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Caron Zlotnick, PhD, Principal Investigator — Women and Infants' Hospital
Locations (4):
- United States (4):
  - New Hope, Attleboro, Massachusetts
  - Battered Women's Shelter of Summit and Medina Counties, Akron, Ohio
  - Center for Women's Behavioral Health at Women and Infants' Hospital, Providence, Rhode Island
  - Sojourner House, Woonsocket, Rhode Island

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SHE Program | Control Condition
Started | 25 | 25
Completed | 21 | 23
Not Completed | 4 | 2
Not completed — Lost to Follow-up | 3 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: NA - patient flow and assignment were as expected.
Groups:
- Total: Total of all reporting groups
Arm/Group | SHE Program | Control Condition | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 24 | 25 | 49
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.3 (11.4) | 35.2 (11.5) | 35.2 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 25 | 50
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 4 | 9
  Not Hispanic or Latino | 20 | 21 | 41
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 11 | 21
  White | 9 | 10 | 19
  More than one race | 1 | 3 | 4
  Unknown or Not Reported | 5 | 0 | 5
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50
% drug using/heavy drinking days [Median (Standard Deviation); unit: % drug using/heavy drinking days] | 0.54 (0.38) | 0.66 (0.38) | 0.59 (0.37)

OUTCOME MEASURES:

1. Primary Outcome: Alcohol and Substance Use: Timeline Follow-back (TLFB)-Modified Computer Version
Description: The computer-based TLFB will assess drug use and heavy drinking (4+ standard drinks) days for the past week and the past 90 days. For primary analysis, days using drugs and heavy drinking days will be combined to create a single variable that reflects the total number of days that women used drugs or had 4+ drinks. The primary outcome is substance use (heavy drinking or drug using) days over a 6 month post shelter period. We are assessing the change of this number from baseline to 3 months post shelter, and from baseline 6 months post shelter.
Time Frame: Assessed at baseline, and at 3 and 6 months post shelter
Measure: Median (Standard Deviation); unit: % days of drug use or heavy drinking
Arm/Group | SHE Program | Control Condition
Number analyzed (Participants) | 25 | 25
% days of drug use or heavy drinking
  Baseline | 0.54 (0.38) | 0.66 (0.38)
  3 months post-shelter | 0.12 (0.38) | 0.29 (0.38)
  6 months post-shelter | 0.21 (0.42) | 0.16 (0.21)
Statistical Analysis 1: Comparison: SHE Program vs Control Condition; Test type: Superiority; p = 0.560, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: SHE Program vs Control Condition; Differences between conditions in the change in % heavy drinking/using days from baseline to 6 months; Test type: Superiority; p = 0.760, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: The Treatment Services Review (TSR)
Description: The Treatment Services Review will be used to assess total times using substance use services (both treatment and self-help utilization) received (including outpatient, day patient, residential treatment, NA, AA) to capture the extent to which women are reaching out to access recovery-related resources. The TSR will assess number of times attending substance use services, divided by the number of days in the reporting period.
Time Frame: Assessed at baseline, and again at 3 and 6 months later
Measure: Median (Standard Deviation); unit: times using substance use services/day
Arm/Group | SHE Program | Control Condition
Number analyzed (Participants) | 25 | 25
times using substance use services/day
  Baseline | 0.00 (0.05) | 0.01 (0.25)
  3 months post-shelter | 0.00 (0.23) | 0.00 (0.22)
  6 months post-shelter | 0.00 (0.22) | 0.00 (0.16)
Statistical Analysis 1: Comparison: SHE Program vs Control Condition; Test type: Superiority; p = 0.026, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: SHE Program vs Control Condition; Distributions were badly skewed, and the sample was too small for ZINB or other analyses. Therefore, we analyzed differences between conditions in changes in services/day over time (i.e., from baseline to 6 month post-shelter follow-up) using the Mann-Whitney U; Test type: Superiority; p = 0.029, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: The Composite Abuse Scale (CAS)
Description: The CAS is a widely used self-report of behaviors scale with 4 subscales that measure severe, combined abuse, emotional abuse, physical abuse, and harassment. The CAS has recently been published in the Centers for Disease Control and Prevention compendium of intimate partner violence measures. It consists of 30 items presented in a six point format requiring respondents to answer "never", "only once", "several times", "monthly", "weekly" or "daily" in a twelve month period. Below we present the CAS victimization scores. Scores range from 0 to 145; higher scores are worse.
Time Frame: Assessed at baseline, and again at 3 and 6 months after shelter release
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SHE Program | Control Condition
Number analyzed (Participants) | 25 | 25
score on a scale
  Baseline | 52.8 (22.6) | 74.4 (40.5)
  3 months post-shelter | 9.4 (11.5) | 17.7 (32.8)
  6 months post-shelter | 14.1 (23.8) | 4.9 (10.6)
Statistical Analysis 1: Comparison: SHE Program vs Control Condition; Test type: Superiority; p = 0.325, Mixed Models Analysis — We used hierarchical linear modeling (HLM) to predict 3-mo and 6-mo post-shelter scores from treatment condition, using baseline score as a covariate; Mean Difference (Final Values) = 4.5, 95% CI 2-sided [-4.5 to 13.5]

4. Secondary Outcome: The Cyber Stalking Scale
Description: The Cyber Stalking Scale measure is a 6 -item measure and assesses the use of technologies in stalking and harassment. Scores range from 0 to 12. Lower is better (indicated less Cyber Stalking).
Time Frame: Assessed at baseline, and again at 3 and 6 months later
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SHE Program | Control Condition
Number analyzed (Participants) | 23 | 23
score on a scale
  Baseline | 9.53 (3.01) | 7.39 (4.29)
  3 months post-shelter | 4.95 (4.54) | 3.30 (4.45)
  6 months post-shelter | 3.89 (4.27) | 2.00 (3.23)
Statistical Analysis 1: Comparison: SHE Program vs Control Condition; Test type: Superiority; p = 0.192, Mixed Models Analysis — We used HLM to predict Cyber-Stalking Scores across 3 and 6 month post shelter follow-up points from treatment condition, using baseline score as a covariate; Mean Difference (Final Values) = 1.19, 95% CI 2-sided [-0.61 to 2.98] — Higher scores represent more cyber-stalking over follow-up

5. Secondary Outcome: Safety Behavior Checklist (SBC)
Description: Safety Behavior Checklist (SBC) has 15 items that assess the use of strategies suggested to keep victim safe (e.g., hiding money and extra clothing). Scores range from 0 to 15; higher scores are better (indicating more safety behaviors used).
Time Frame: Assessed at baseline, and again at 3 and 6 months after shelter release
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SHE Program | Control Condition
Number analyzed (Participants) | 25 | 25
score on a scale
  Baseline | 7.3 (2.7) | 7.3 (4.0)
  3 months post-shelter | 4.5 (3.4) | 5.7 (4.9)
  6 months post-shelter | 2.8 (3.8) | 4.9 (5.3)
Statistical Analysis 1: Comparison: SHE Program vs Control Condition; Test type: Superiority; p = 0.119, Mixed Models Analysis — We conducted HLM predicting SBC Total scores at 3 and 6 months post-shelter release from treatment condition, using baseline SBC score as a covariate; Mean Difference (Final Values) = -1.43, 95% CI 2-sided [-3.24 to 0.38] — Higher is better (reflecting more safety behaviors used)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from baseline to 6 months after the participant left the shelter--varies from 6 months to 1 1/2 years depending on the participant.
Description: In addition, the DSMB also included possible partner violence due to a child welfare report made by study participant and/or study staff (if have children) during the duration of the study.
Arm/Group | SHE Program | Control Condition
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 15/25 | 16/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SHE Program (N=25) | Control Condition (N=25)
Hospitalization-general medical issue (Surgical and medical procedures) | 3 (3) | 3 (3)
Hospitalization-IPV related (Injury, poisoning and procedural complications) | 4 (4) | 7 (7)
Hospitalization-inpatient-psyc (Psychiatric disorders) | 5 (8) | 5 (16)
IPV-sought no medical care (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
IPV-emergency room visit only (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-03-15): https://cdn.clinicaltrials.gov/large-docs/33/NCT02629133/SAP_002.pdf
  • Study Protocol (2017-03-15): https://cdn.clinicaltrials.gov/large-docs/33/NCT02629133/Prot_003.pdf